CLINICAL TRIAL: NCT01075620
Title: Comparison of Nonposterior- and Posterior-Stabilized Mobile-Bearing Total Knee Arthroplasty A Prospective, Randomized Study
Brief Title: Comparison of Nonposterior- and Posterior-Stabilized Mobile-Bearing Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Young-Hoo, Kim M.D. Professor, Ewha Womans University Mokdong Hospital Joint Replacement Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-2-16
Record Dates: First submitted 2010-02-16; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-01

CONDITIONS: Osteoarthritis
Keywords: rotating platform; posterior stabilized; non-posterior stabilized
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PFC sigma RP (Experimental): Posterior stabilized rotating platform knee (press Fit Condylar Sigma rotating-platform, Depuy, Warsaw, Indiana)
  Interventions: Device: PFC-Sigma RP
- LCS RP (Active Comparator): non posterior stabilized Low Contact Stress Rotating-Platform; Depuy, Warsaw, Indiana
  Interventions: Device: LPS RP

INTERVENTIONS:
Device: PFC-Sigma RP — Posterior stabilizing rotating platform total knee components
  Other Names: PFC sigma RP
  Arms: PFC sigma RP
Device: LPS RP — non-posterior stabilized rotating platform design
  Other Names: LCS RP
  Arms: LCS RP

SUMMARY:
The purpose of this study is to determine if there are any clinical or radiographic differences in non-posterior stabilized rotating mobile bearing design versus a posterior stabilized rotating mobile bearing designs.

DETAILED DESCRIPTION:
Out comes measures were to determine

1. whether the knee and function scores and the radiographic results of the knees with a PFC Sigma RP knee prosthesis would be better than those with an LCS RP prosthesis.
2. whether the patients with a PFC RP knee prosthesis would have a better range of knee motion than those with an LCS RP prosthesis.
3. whether patient satisfaction and preference would be better in the patients having a PFC Sigma RP knee prosthesis than those of patients having an LCS RP knee prosthesis
4. whether complication rate would be less in the knees with a PFC sigma RP knee prosthesis than in the knees with an LCS RP prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* End-stage osteoarthritis of the knee joint requiring total knee arthroplasty with bilateral disease

Exclusion Criteria:

* Inflammatory disease
* patient with other Lower extremity disease which may affect functional outcome
* Neurologic disease effecting patients lower extremity
* Revision surgery
* Patient not medically cleared for bilateral surgery

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2002-05; Primary Completion 2002-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Knee Society knee score | at 3 months, 1 year, than annually

SECONDARY OUTCOMES:
Range of motion | at 3 months, 1 year, than annually

CONTACTS AND LOCATIONS:
Overall Officials: Yoowang Choi, MD, Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea